CLINICAL TRIAL: NCT02107508
Title: The Relationship Between Activity Energy Expenditure and Body Composition in School-age Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huijuan Ruan (Other)
Responsible Party: Sponsor-Investigator, Huijuan Ruan, M.D., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: XHEC-C-2013-021
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Childhood Obesity
Keywords: activity energy expenditure; body composition
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity is increasing rapidly all over the world not only in adults but also among children. As a modifiable component of total energy expenditure (TEE) ,the amount of energy expended during physical activity plays an important role in preventing weight gain. Decreased physical activity, coupled with an over-consumption of calories, lead to the change of body composition by storing energy as fat.Although several studies have simultaneously examined body composition with energy expenditure the independent roles of body composition with activity energy expenditure (AEE) are less firmly established. It's suspected shrewdly that energy expenditure is partly influenced by the body composition. The aim of the study is to examine the relation of AEE with body composition in a population of school-age children.

DETAILED DESCRIPTION:
Body composition (ie. FAT% and FFM) will be evaluated by means of bioelectrical impedance analysis (BIA) with Inbody 720 (Biospace, Seoul, South Korea). Anthropometric dimensions will be recorded for all participants according to standard procedures. Height will be recorded to the nearest 1.0mm by using a field stadiometer (Seca Corporation, Germany). FitMate metabolic system (Cosmed, Rome, Italy) will be used to estimate AEE. Subjects will be tested in a 10-minute submaximal exercise test using the FitMate systems while taking cycling test at 50 Watts on an electrically braked bicycle ergometer. Each subject will be connected to a calibrated respiratory gas analyzer, a portable metabolic analyzer designed for measurement of oxygen consumption during exercise via a face mask. Heart rate will be simultaneously measured with the use of a Cosmed wireless HR monitor to track the participant's heart rate level.

ELIGIBILITY:
Inclusion Criteria:

* Children in Shanghai

Exclusion Criteria:

* cardiovascular disease
* asthma
* severe disease conditions such as cancer and renal failure
* taking steroids (corticosteroids) or antidepressants

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children in Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
body composition | up to 30 days after participating in the study
  Each participant will be weighted while wearing light clothing, after fasting for at least 4 hours and emptying the bladder. Body composition, such as body weight, fat mass(FM), fat percentage (FAT%) and free fat mass (FFM) will be measured by bioelectrical impedance analysis(BIA) with Inbody 720 (Biospace, Seoul, South Korea).Body composition measurement will be compared between the normal weight group and overweight/obesity group.

SECONDARY OUTCOMES:
activity energy expenditure (AEE) | up to 30 days after participating in the study
  Each participant will be asked to perform a cycling test to measure the AEE. Measurements will be recorded in the early afternoon. Total AEE (kcal) will be measured in the test. The exercise time will be adjusted by using the AEE (kcal/min), which was calculated as Total AEE/min. The weight-adjusted AEE (kcal/kg/min) will be calculated to facilitate comparisons between persons. AEE will be compared between the overweight/obesity group and normal weight group.

CONTACTS AND LOCATIONS:
Overall Officials: Qingya Tang, M.D., Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China